CLINICAL TRIAL: NCT01678053
Title: A Randomized Controlled Trial Comparing Proton Pump Inhibitor Therapy With and Without Interarytenoid Botulinum Toxin Injection for Vocal Fold Granuloma
Brief Title: Efficacy Study of Botulinum Toxin (BOTOX) Injections to Treat Vocal Fold Granulomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Was not able to recruit patients for randomization.
Sponsor: Phillip Song, MD (Other)
Responsible Party: Sponsor-Investigator, Phillip Song, MD, Otolaryngologist, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-090H
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Contact Ulcer of Vocal Folds; Granuloma of Vocal Cords; Granuloma, Laryngeal; Granuloma
Keywords: Botulinum Toxins, Type A
MeSH Terms: conditions — Granuloma, Laryngeal; Granuloma | interventions — Botulinum Toxins, Type A; Omeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPI and BOTOX (Experimental): onabotulinumtoxinA (BOTOX), injection, 10 units, one time; omeprazole 40mg po bid (standard of care) for 3 months
  Interventions: Drug: onabotulinumtoxinA; Drug: omeprazole (proton pump inhibitor)
- Proton pump inhibitor only (Other): omeprazole 40mg po bid for 3 months(standard of care)
  Interventions: Drug: omeprazole (proton pump inhibitor)

INTERVENTIONS:
Drug: onabotulinumtoxinA — Botulinum toxin A is injected into the larynx in order to treat vocal fold granulomas.
  Other Names: BOTOX; Botulinum toxin A
  Arms: PPI and BOTOX
Drug: omeprazole (proton pump inhibitor) — Standard therapy of anti-reflux medications using omeprazole or equivalent PPI.
  Other Names: omeprazole

SUMMARY:
Vocal process granulomas are inflammatory masses caused in part by vocal trauma that arise in the posterior aspect of the vocal folds and result in throat pain, difficulty swallowing, hoarseness, and globus sensation. Antireflux therapy treats most granulomas, but many are recalcitrant to this therapy or take months to years to resolve. Botulinum toxin injection into the thyroarytenoid muscle has been effectively employed for recalcitrant granuloma, but causes significant voice loss, occasional difficulty swallowing and, in our clinical experience, is associated with significant recurrence. The investigators propose injecting another muscle in the larynx called the interarytenoid muscle with botulinum toxin type A to maintain the benefit of injection with less loss of voice. The investigators have shown the effectiveness of this treatment in a small, retrospective analysis.

DETAILED DESCRIPTION:
Vocal fold granulomas may be due to reflux, voice trauma, intubation, multiple or unknown etiologies. Regimens of voice therapy and anti-reflux medications have show resolution rates varying from 38% to 100%, with recurrence rates of 15-20%, and up to 50-92% in surgical-operated on recalcitrant granulomas. Nasri and colleagues first proposed thyroarytenoid botulinum toxin type A (BOTOX) injections for vocal fold granulomas with success. They posited that the chemically paralyzed muscle would result in limited contact at the site of the granuloma, allowing for healing. Damrose and Damrose further showed that thyroarytenoid BOTOX injections were effective in treating recalcitrant vocal fold granulomas. Both of the above groups noted hoarseness as an expected side effect. Pham and colleagues showed complete resolution of granulomas in 2-8 weeks after treatment with thyroarytenoid BOTOX injections. This was compared to mean granuloma resolution of 5.7 months proton pump inhibitor therapy alone. The investigators reviewed eight patients treated for recalcitrant vocal fold granuloma at Mass Eye and Ear with interarytenoid BOTOX injections and found no serious adverse effects and complete response in seven cases. The investigators now seek to compare interarytenoid BOTOX injections to standard anti-reflux therapy alone to see if the addition of IA Botox injections improves response rates at 3 months. The investigators chose this timeframe since 86% of granulomas treated in our retrospective study had resolved 3 months after initiation of treatment compared to 25% of granulomas treated with medical management.

The investigators will not include a Thyroarytenoid injection arm in this study as this technique has not been useful in our clinical experience.

For those who consent, a Voice Handicap Index survey (6 - see attached) will be completed. Participants will then be randomized to undergo only medical therapy with omeprazole (40mg by mouth twice daily ) or an interarytenoid BOTOX injection followed by the same reflux regimen. Randomization will be performed by the Tufts online randomization plan, which may be found at: http://www.tufts.edu/~gdallal/PLANDOC.HTM. This program generates a random order in which participants will be enrolled in either of the two arms of the study.

The injection will consist of 10 units of botulinum toxin injected into the interarytenoid muscle under fiberoptic visualization. All participants will remain on the PPI therapy for the duration of the study. Participants will receive prescriptions for PPI medication from the attending Laryngologist and participants will then be responsible for acquiring and taking their medications.

Injections will be performed per standard MEEI Laryngology protocol for interarytenoid BOTOX injection. Participants will then be evaluated at 1.5 months, 3 months and 6 months with fiberoptic examination as well as Voice Handicap Index & Reflux Symptom Index. Participants in the medication only arm who continue to have a granuloma at 3 months will receive a BOTOX injection. They will be re-evaluated 3 months after the injection. Examinations will be recorded and reviewed by blinded reviewers.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 years old and older with vocal fold granulomas
* willing to attend all follow-up appointments

Exclusion Criteria:

* pregnant females
* woman who are nursing
* minors and other patients unable to give informed consent
* patients taking Plavix
* patients with:
* impaired laryngeal motion as the result of neurological impairment
* vocal fold immobility
* pre-existing oropharyngeal swallowing problems
* history of radiation therapy
* history of aspiration pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Complete resolution of vocal fold granuloma | 3 months

SECONDARY OUTCOMES:
Voice Handicap Index score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Song, M.D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Background] de Lima Pontes PA, De Biase NG, Gadelha EC. Clinical evolution of laryngeal granulomas: treatment and prognosis. Laryngoscope. 1999 Feb;109(2 Pt 1):289-94. doi: 10.1097/00005537-199902000-00021. PMID 10890781
- [Background] Emami AJ, Morrison M, Rammage L, Bosch D. Treatment of laryngeal contact ulcers and granulomas: a 12-year retrospective analysis. J Voice. 1999 Dec;13(4):612-7. doi: 10.1016/s0892-1997(99)80015-0. PMID 10622526
- [Background] Pham J, Yin S, Morgan M, Stucker F, Nathan CO. Botulinum toxin: helpful adjunct to early resolution of laryngeal granulomas. J Laryngol Otol. 2004 Oct;118(10):781-5. doi: 10.1258/0022215042450788. PMID 15550184
- [Background] Nasri S, Sercarz JA, McAlpin T, Berke GS. Treatment of vocal fold granuloma using botulinum toxin type A. Laryngoscope. 1995 Jun;105(6):585-8. doi: 10.1288/00005537-199506000-00005. PMID 7769940
- [Background] Damrose EJ, Damrose JF. Botulinum toxin as adjunctive therapy in refractory laryngeal granuloma. J Laryngol Otol. 2008 Aug;122(8):824-8. doi: 10.1017/S0022215107000710. Epub 2007 Oct 2. PMID 17908354
- [Background] Ylitalo R, Lindestad PA. A retrospective study of contact granuloma. Laryngoscope. 1999 Mar;109(3):433-6. doi: 10.1097/00005537-199903000-00017. PMID 10089971